CLINICAL TRIAL: NCT07247006
Title: Ketamine-Assisted Psychotherapy for Treatment-Resistant Depression
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Paul Geha, Associate Professor - Department of Psychiatry, Research (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010828
Record Dates: First submitted 2025-11-06; First posted 2025-11-25 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Treatment Resistant Depression (TRD); Chronic Pain
Keywords: depression; fmri
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Chronic Pain; Depression | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TRD group (Experimental)
  Interventions: Drug: Ketamine hydrochloride injection

INTERVENTIONS:
Drug: Ketamine hydrochloride injection — 0.5-1mg/kg intramuscular (IM) injection of ketamine
  Other Names: ketamine; ketalar

SUMMARY:
The goal of this clinical trial is to understand the effect of ketamine on the brain in people with treatment-resistant depression (TRD). TRD occurs in around a third of people with depression and leads to higher suicide rates compared to those with major depressive disorder. A desperate need for a rapid acting antidepressant drug (RAAD) is needed to help improve quality of life for people with TRD. Ketamine has been shown to be a RAAD, and esketamine (a form of ketamine) was approved by the FDA to treat TRD. Ketamine has been known to cause dissociative experiences, that can lead to an increase in the "Openness to Experience" personality trait and psychological flexibility that occurs at "peak experience". This has been shown to improve mental health conditions and lower suicide risk. This study aims to further understand if there is a connection between this new change of mind and changes in brain activity. Ketamine has been shown to improve brain plasticity as well, specifically in the frontolimbic region of the brain, an area associated with depression. The investigators are analyzing the brain using functional magnetic resonance imaging (fMRI), a method used to measure brain activity. The frontolimbic region is also associated with cognitive flexibility and emotional processing, an important hurdle in treating TRD. Due to this, the investigators are pairing the ketamine treatment with psychotherapy sessions, to guide the processing experience, which can lead to higher emotional flexibility.

The main questions this study aims to answer are:

* Are frontolimibic plasticity circuitry changes associated with openness to experience and peak experience?
* Is it feasible to recruit and retain people through a two-month KAP study?
* Is the structure of the study effective for treating TRD?

Participants will:

* Visit the facilities 6-8 times
* Complete 2 MRI brain scans
* Complete 3-4 psychotherapy sessions
* Receive 1-2 doses of ketamine
* Complete online surveys between 3-4 visits

DETAILED DESCRIPTION:
The proposed study is a single center study investigating the effect of ketamine modulation on the brain signature of treatment resistant depression (TRD). The patients will undergo 2 scanning visits (baseline and follow-up). They will also receive 1-2 treatments of ketamine IM injection and 3-4 psychotherapy sessions.

Patients with TRD will be asked to come to the PI's lab for 2 visits, and 6 in the Department of Psychiatry. On visit 1, after consenting and doing the drug screen, the subjects will be asked questions on their depression experience. Subjects will then fill out demographic and clinical questionnaire to assess mood, anxiety, pain, history of early trauma, and stress. Patients will be asked to rate their depression and pain level using a visual analogue scale (VAS).

During visit 1, Drs. Geha and Swogger will interview the patients to inquire about any prior drug allergies including allergies to medications that could be possibly used in this study (ketamine/ondansetron/lorazepam/clonidine). Possible side effects will be explained to the patients. They will then undergo 60 minutes of functional and structural brain scanning, which will serve as a baseline scan.

Visits 2 and 3 will be psychotherapy sessions with Dr. Swogger to prepare for the ketamine session and focus on their difficulties and goals for the medicine session. Strategies for working with ketamine will be reviewed.

Visits 4 and 6 will be the ketamine IM injection sessions. Visit 4 they will receive 0.5 mg/kg but will not exceed 60 mg regardless of weight. Visit 6 may be a higher dose, but will not exceed 60 mg. The dose will be determined by Drs. Geha and Swogger based on the patients' experience and response in visit 4. Ondansetron will be available for nausea, lorazepam for uncontrolled agitation, and clonidine for uncontrolled hypertension. Throughout the visits members of the study team will be present to ensure patient comfort and offer reassurance, redirection, etc. They will also take notes for later processing in psychotherapy visits. When the patient emerges from non-ordinary state of consciousness, they will complete the MEQ, and the study team will complete CADSS-6 and record any other pertinent information about the experience. Once it is deemed safe, the patient may leave via someone driving them home after the visit and will be instructed on safety measures for the rest of the day.

Visits 5 and 7 will be follow up psychotherapy visits the day after the ketamine treatment. They will discuss and process the experience. If the patient wishes not to receive another dosage, then visit 7 will not occur and they will proceed with visit 8 after visit 5.

Visit 8 is conducted in the PI's lab about 4 weeks after visit 5 (one dose) or 7 (two doses). This will include answering similar questionnaires from the baseline visit to assess depression, pain, anxiety, mood, trauma, and personality. The patient will discuss the accessibility and feasibility of the study with Dr. Swogger or a member of the study team. Then they will conduct a follow up functional and structural brain imagining scan, lasting for 60 minutes.

For 7 days after visit 1, 7 days after each ketamine session, and 7 days before visit 8, the patient will complete quick at home surveys to assess depression and pain.

Throughout the study the investigators will assess depression, mood, pain, and Openness to Experience using the questionnaires below:

* Hamilton Depression Rating Scale (HDRS or HAM-D): Clinical tool that assesses the severity of depression. Includes 17 questions that assess depressed mood, suicidal ideation, anxiety, and somatic symptoms.
* Beck Depression Inventory (BDI): A 21-item questionnaire that measures depression. It is not used to diagnose, but to monitor presence and severity of symptoms and for monitoring treatment.
* NEO Five-Factor Inventory (NEO-FFI): Personality assessment tool to measure the personality domains of Neuroticism, Extraversion, Openness to Experience, Agreeableness, and Conscientiousness.
* The McGill Pain Questionnaire - Short Form 2 (SF-MPQ-2): A self-reporting measure of pain used to assess quality and intensity of pain qualitatively. This version includes neuropathic and non-neuropathic pain conditions with a total of 22 items, with response options of 0-10, with 0 being no pain, and 10 being the worst imaginable pain.
* Numerical Pain Scale (NRS): A simple used to assess pain intensity where the subject rates their pain on a scale of 0 to 10, 10 being the worst possible pain.
* Visual Analog Scale (VAS): A tool used to assess pain intensity, with a line with one end labeled 0 (no pain) and 100 (worst pain possible) and subjects place the curser where they would rate their current pain intensity. The curser is not labeled with a number as it is moved. There will also be one for depression (no depression symptoms to worst depression imaginable).
* Beck Anxiety Inventory (BAI): A self-report questionnaire that assesses the severity and frequency of anxiety symptoms. It is a 21-item questionnaire with answer options going 0-3, with 0 being no effect on the individual and 3 being severely bothersome.
* Childhood & Recent Traumatic Events Scale (CTES): A psychological tool to measures past and recent trauma. The childhood portion focuses on trauma that occurred before the age of 17. The recent events portion assesses trauma that occurred in the last 3 years. They both ask about death of a family member, sexual trauma, violence, and severe illness/injury. Additionally, the childhood portion asks about parental separation, while the recent events portion asks about spousal separation.
* Modified Antidepressant Treatment History Form (ATHF): A widely used instrument that provides objective criteria to make an assessment if an antidepressant treatment was a failed trial or adequate trial, helping to confirm treatment resistant depression. The investigators will also be asking about previous psychotherapy treatments.

The trial acceptability and ketamine experience will be assessed using the questionnaires below:

* Mystical Experiences Questionnaire: A questionnaire that is comprised of 30 items and provides systematic and empirical methods of assessing feelings of unity, transcendence, and altered states of consciousness after taking a psychedelic. It was originally designed for psilocybin treatments; therefore, the questionnaire will have the word "psilocybin" replaced by "ketamine" to better fit this study.
* Clinician Administered Dissociative States Scales (CADSS-6): Short form version of CADSS, with only 6 items. It is designed to measure dissociative symptoms, and it has been utilized by many clinical trials featuring ketamine.
* Ketamine Side Effect Tool (KSET): A form that is used clinically and in research to assess side effects that occur with ketamine treatment.
* NIH Stroke Scale Neurological Assessment Flow Sheet: A set of neurological checks to assess patient level of consciousness and alertness.
* Likert Scale for Acceptability: A measure of acceptability for the study. It will be used as a feedback form and to help measure feasibility for the study.

ELIGIBILITY:
Inclusion Criteria

The following inclusion criteria must be met for all subjects to be considered eligible to participate:

1. 18 years old or older
2. Able to speak, read, and understand English
3. In generally stable health
4. Must have treatment resistant depression, as defined as scoring in the moderate or above range on the HDRS and having failed two adequate trials of antidepressants in the last two years.

Exclusion Criteria

General exclusion criteria for all subjects include:

1. Uncontrolled hypertension
2. Impaired cardiac status

   a. Abnormal ECG report in the last month prior to screening
3. Chronic Obstructive Pulmonary Disease
4. Congenital Long QT Syndrome
5. ≥265lbs or 120kg
6. Severe obesity (BMI ≥40)
7. Increased intracranial or cerebrospinal pressure
8. Pregnancy or breastfeeding
9. Hyperthyroidism
10. Prior adverse response to ketamine, including allergic reaction
11. Symptoms of psychosis or prodromal phase
12. Severe personality disorder
13. Autistic Spectrum Disorders
14. Bipolar disorder
15. History of substance abuse, defined as a score of three or more on Drug Abuse scale (prior use of psychedelics allowed)
16. Past-year suicide attempt or ongoing ideation with intent to act
17. All exclusion criteria for magnetic resonance imaging safety: any metallic implants, brain or skull abnormalities, tattoos on large body parts, and claustrophobia.
18. Taking medications that could interact with ketamine. Examples include but are not limited to: any types of stimulants, aripiprazole, diphenhydramine, hydromorphone, escitalopram, fluoxetine, alprazolam, and sertraline. Each subject's current medications will be evaluated for interactions with ketamine before admission into the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Retained in Study Through 2-Month Follow-Up | 2 months post-enrollment
  Retention will be assessed as completion of all scheduled study assessments through the 2-month follow-up. A single value is derived for each participant, coded as 1 (retained) or 0 (not retained). Higher values indicate successful retention; lower values indicate dropout.
Mean Change in Hamilton Depression Rating Scale (HDRS) Total Score | Baseline, once a day for up to 7 days after baseline, within 90 minutes after ketamine dosing session, once a day for up to 7 days after ketamine dosing session, once a day up to 7 days before 2-month follow-up, and at 2-month follow-up
  Depression severity will be measured using the 17-item HDRS (items scored 0-2 or 0-4; total score range 0-52). A single value is derived by summing item scores. Higher scores indicate greater depression severity (worsening); lower scores indicate reduced severity (improvement). Mean change is calculated as post-treatment score minus baseline score.

SECONDARY OUTCOMES:
Mean Change in Numerical Pain Rating Scale Score | Baseline, once a day for up to 7 days after baseline, within 90 minutes after ketamine dosing session, once a day for up to 7 days after ketamine dosing session, once a day up to 7 days before 2-month follow-up, and at 2-month follow-up
  Pain intensity will be assessed using an 11-point Numeric Rating Scale (0 = no pain, 10 = worst imaginable pain). A single value is derived by averaging participant ratings at each time point. Higher scores indicate worse pain; lower scores indicate reduced pain. Mean change is calculated as follow-up score minus baseline score.
Mean Change in NEO Five-Factor Inventory-3 (NEO-FFI-3) Openness Subscale Score | Baseline and 2-month follow-up.
  Openness will be measured using the NEO-FFI-3 Openness subscale (12 items scored 0-4; total score range 0-48). A single value is derived by summing the 12 item scores. Higher scores indicate greater openness; lower scores indicate reduced openness. Mean change is calculated as follow-up score minus baseline score.
Mean Acceptability Rating of Ketamine-Assisted Psychotherapy | At 2 month follow-up
  Acceptability will be assessed using a 5-point Likert scale (1 = low acceptability, 5 = high acceptability). A single value is derived by averaging scores across participants. Higher scores indicate greater acceptability; lower scores indicate lower acceptability.
Proportion of Participants Reporting Adverse Events (AEs) | Throughout the 8-week study.
  Adverse events will be graded using the Common Terminology Criteria for Adverse Events (CTCAE v5.0; 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = fatal). A single value is derived for each participant as the highest AE grade experienced. Higher values indicate more severe AEs; lower values indicate milder or no AEs.

OTHER OUTCOMES:
Mean Mystical Experience Questionnaire (MEQ-30) Total Score | within 1-2 days after each ketamine dosing session
  Mystical experiences will be measured using the MEQ-30 (30 items scored 0-5; total score range 0-150). A single value is derived by summing item scores. Higher scores indicate more intense mystical experiences; lower scores indicate fewer or weaker mystical experiences.
8. Mean Change in Resting-State fMRI Whole Brain Functional Connectivity | Baseline and at 2 month follow-up
  Functional connectivity will be measured using resting-state fMRI. Correlations between 400 cortical ROIs (Schaefer atlas) and subcortical ROIs (Harvard-Oxford atlas) will be calculated. A single value per participant is derived as the mean Fisher-Z transformed correlation coefficient across all ROI pairs. Higher values indicate stronger connectivity; lower values indicate weaker connectivity. Mean change is calculated as post-treatment value minus baseline value.
Mean Change in Subcortical Brain Volume | Baseline and at 2 month follow up
  Volumes of subcortical structures will be calculated from MRI scans using FSL-FIRST and FreeSurfer. A single value per participant is derived by summing the volumes of predefined structures (mm³). Higher values indicate larger volumes; lower values indicate smaller volumes. Mean change is calculated as post-treatment volume minus baseline volume.
Clinician-Administered Dissociative States Scale (CADSS-6) Total Score | within 90 minutes after each ketamine dosing session
  Dissociation will be measured using the CADSS-6 (6 items scored 0-4; total score range 0-24). A single value is derived by summing item scores. Higher scores indicate greater dissociation; lower scores indicate less dissociation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No